CLINICAL TRIAL: NCT05445453
Title: Museum Prescription by a Physician for a Visit to the Montreal Museum of Fine Arts: Assessment of Effects.
Brief Title: Museum Prescription by a Physician for a Visit to the MBAM
Acronym: PM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal (Other Government)
Responsible Party: Principal Investigator, Olivier Beauchet, MD, PhD, Senior researcher, Director of laboratory, Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MP-53-2023-2627
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Quality of Life; Social Isolation
Keywords: Arts; Well-being; Mental Health
MeSH Terms: conditions — Social Isolation; Arts syndrome; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This study is experimental, prospective, open-label, non-randomized, pre-post intervention with a single group of participants who will be their own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Physicians participating in the research project will be able to prescribe a visit to the Museum to any of their patients for whom they deem this museum prescription necessary. Only patients who meet the inclusion criteria will be offered to participate in the research.
  If patients refuse or do not meet the inclusion criteria, they may be prescribed a museum visit but will not be offered the study.
  After obtaining informed consent, the patient will be asked to complete 2 sets of self-administered questionnaires: in the 2 days prior to the visit and in the 2 days following the MBAM visit.
  Interventions: Other: Museum visit

INTERVENTIONS:
Other: Museum visit — The intervention is a visit of the MMFA. This visit can be done alone or accompanied.
  The visit of the MMFA is free for the patient.

SUMMARY:
In recent years, museums have participated in the patient care journey by using art to enhance their quality of life and well-being. Since 2015, the Montreal Museum of Fine Arts (MMFA) and Dr. Beauchet have developed an Action-Research program exploring the effects of participatory art activities for community elders conducted at the MMFA, known as the Arts & Longevity Lab (ALL). The mandate of ALL is to improve the well-being, quality of life and health (i.e. mental and physical state) of individuals and patients through the practice of visual arts activities (i.e. arts that produce objects perceived by the eyes).

Since 2019, the MMFA has developed in collaboration with Médecins Francophones du Canada museum visits prescribed by a primary care physician as a new intervention. Today, it is necessary to improve the knowledge on the effects of this museum visit prescription

The overall objective of this study is to examine the effects of a visit to the MMFA prescribed by a primary care physician on the mental health (well-being and quality of life) of patients living in Montreal.

ELIGIBILITY:
Inclusion Criteria:

* age 18 and over
* having Internet access at home with an electronic device (computer, keyboard, or smartphone)
* having no dementia
* speaking English or French
* committing to visiting the museum within 3 months of the prescription.

Exclusion Criteria:

* individuals participating in a clinical trial at the same time, to avoid interference with the results of the intervention being studied in this protocol
* individuals with dementia. There are no tests for dementia. The physicians involved in the pre-recruitment process are aware of the cognitive status of their patients. Therefore, they will be able to avoid offering the study to a patient with dementia if such a diagnosis appears in the medical file.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Quality of life | 3 months
  Quality of life will be assessed using the EuroQol-5D (EQ-5D).
  EuroQol-5D is composed of two parts:
  * a five-question questionnaire with a score per question ranging from 1 (no problem) to 5 (severe problem), so that the sum ranged from 0 (no problem) to 25 (severe problem).
  * a visual analogue scale on participants' perceived health. This scale is numbered from 0 (i.e., the worst health the participant can imagine) to 100 (i.e., the best health the participant can imagine).
  This questionnaire will be completed online on the CRIUGM web platform using an electronic device.
Well-being | 3 months
  Well-being will be assessed using the Warwick-Edinburgh Mental Well-being Scale (WEMWBS).
  The WEMWBS is a validated questionnaire composed by a 14-item positively worded scale and five response categories. It covers most aspects of positive mental health (positive thoughts and feelings).
  This questionnaire will be completed online on the CRIUGM web platform using an electronic device.

SECONDARY OUTCOMES:
Physical Health Status | 3 months
  Physical health status will be assessed using the CRIUGM Self-AdMinistered questionnaire (CESAM).
  The CESAM has been previously developed and validated.
  It is composed of 20 items exploring several domains:
  * weight loss and its extent;
  * polypharmacy defined by a number of therapeutic classes taken on a daily basis ≥ 5;
  * vision, hearing, and memory problems;
  * use of home support;
  * 6-item activities of daily living scale, 4-item instrumental activities of daily living scale;
  * mood assessed
  * regular physical activity defined as at least 1 hour per week in the past month;
  * and history of falls in the past 12 months.
  The CESAM provides two complementary scores:
  1. An overall frailty score ranging from 0 to 18
  2. A four-stage categorization of frailty
  This questionnaire will be completed online on the CRIUGM web platform using an electronic device.
Social Isolation | 3 months
  Social isolation will be assessed using the 11-item Duke Social Support Index (DSSI).
  This index includes two subscales:
  * social interaction (i.e., frequency of interactions)
  * subjective support (i.e., satisfaction with emotional support provided).
  The DSSI score ranges from 11 to 33, with higher scores indicating higher levels of social inclusion. Scores for the 11 items are combined and categorized as low (score ≤26), high (score 27-29), and very high (score 30-33). We will use the mean score of the 11-item DSSI and its breakdown into three categories as the primary outcome.
  This questionnaire will be completed online on the CRIUGM web platform using an electronic device.
Prescribing context | 3 months
  Researchers will also study the prescribing context. A document will be filled by primary care physicians to give additional informations on the prescribing context such as the date of the prescription and the reason of the prescription.
Satisfaction from the visit to the museum | 3 months
  A short questionnaire will be given to participants to the intervention at the end of the visit to the museum. This questionnaire will give additionnal information on the satisfaction from the visit and whether the visit was made alone or accompanied.

CONTACTS AND LOCATIONS:
Locations (1):
- CRIUGM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beauchet O, Moret A, Deveault M, Thiboutot C, Parent N, Boyer H, Galery K. Physician-prescribed museum visit benefits on mental health: results of an experimental study. Front Med (Lausanne). 2025 May 14;12:1590145. doi: 10.3389/fmed.2025.1590145. eCollection 2025. PMID 40438362